CLINICAL TRIAL: NCT06137235
Title: A Randomized, Controlled, Double-blind Parallel Group Trial to Study the Effects of an Infant Formula and a follow-on Formula Containing Bio-active Ingredients on Growth, Tolerance and Infections in Healthy Term Infants
Brief Title: Effects of an Infant Formula and follow-on Formula Containing Bio-active Ingredients on Growth, Tolerance and Infections
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: Armadillo
Record Dates: First submitted 2023-11-14; First posted 2023-11-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Growth; Infections
Keywords: infant nutrition; growth; gut comfort; product tolerance; infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- test formula (Experimental): infant formula and follow-on formula with bioactive ingredients
  Interventions: Other: cows milk infant formula and follow-on formula with bioactive ingredients
- control formula (Active Comparator): standard infant formula and follow-on formula
  Interventions: Other: standard cows milk infant formula and follow-on formula

INTERVENTIONS:
Other: cows milk infant formula and follow-on formula with bioactive ingredients — infant formula and follow-on formula with bioactive ingredients
  Arms: test formula
Other: standard cows milk infant formula and follow-on formula — standard cows milk infant formula and follow-on formula
  Arms: control formula

SUMMARY:
In this clinical trial, the growth (weight for age), product tolerance (product intake, comfort) and infection-related symptoms of healthy infants consuming an IF and FOF containing bio-active ingredients will be evaluated and compared to a group of infants consuming a standard IF and FOF.

DETAILED DESCRIPTION:
In this clinical trial, the growth (weight for age), product tolerance (product intake, comfort) and infection-related symptoms of healthy infants consuming an IF and FOF containing bio-active ingredients will be evaluated and compared to a group of infants consuming a standard IF and FOF, until the age of 1y. 456 healthy term infants who are exclusively formula-fed will be included <2mo of age. An exploratory follow-up assessment will be done at the age of 2 and 3 years to study sustained health effects.

ELIGIBILITY:
Inclusion Criteria:

* Full-term infants
* Healthy birthweight: 2500 g ≤ birthweight ≤ 4200 g
* Boys and girls
* Apparently healthy at birth and screening
* Weight-for-age Z-score (WAZ) at screening within the normal range according to WHO Child Growth Standards
* Age at enrolment: ≤60 days of age
* If age at inclusion ≤1 month: infants exclusively formula fed for at least 5 days prior to inclusion
* If 1 month < age at inclusion ≤ 2 months: infants exclusively formula fed since 1 month old2
* Being available for follow up until the age of 12 months
* Written informed consent from parent(s) and/or legal guardian(s) aged ≥18 years

Exclusion Criteria:

* Severe acquired or congenital diseases, mental or physical disorders, including cow's milk protein allergy (CMA), lactose intolerance and diagnosed medical conditions that are known to affect study outcomes (e.g. functional gastro-intestinal disorders (FGID))
* Incapability of parents to comply with the study protocol
* Illiterate parents (i.e. not able to read and write in local language)
* Participation in another clinical trial
* Unwillingness to accept the formula supplied by the study as the only formula for their child until the age of 12 months
* Infants fed a special diet other than standard cow's or goat's milk based (non-hydrolyzed) infant formula prior to inclusion

Ages: 5 Days to 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 456 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
weight | until age of 6 months
  weight for age, compared to WHO growth curve, for test group only
infection-related morbidity episodes, parent-reported | 6 - 12 months of age
  number of parental-reported respiratory and gut infection-related symptoms, compared between test and control group

SECONDARY OUTCOMES:
weight | until the age of 6 months
  weight for age, compared to WHO growth curve, for control group
length | until the age of 6 months
  length in cm
head circumference | until the age of 6 months
  head circumference in cm
BMI | until the age of 6 months
  BMI in kg/m2
product tolerance: GI comfort | until the age of 6 months
  GI comfort questionnaire
product tolerance: stool frequency and consistency | until the age of 6 months
  stool frequency and consistency questionnaire
product tolerance: product intake | until the age of 6 months
  product intake (ml/feeding, ml/day)
Duration of infection-related episodes | 6 - 12 months of age
  duration of parental-reported respiratory and gut infection-related symptoms in summed days
infection-related morbidity episodes, physician-diagnosed | 6 - 12 months of age
  number of physician-diagnosed respiratory and gut infection-related symptoms

OTHER OUTCOMES:
weight | at the age of 2 and 3 years
  weight in kg
length | at the age of 2 and 3 years
  length in m
head circumference | at the age of 2 and 3 years
  head circumference in cm
BMI | at the age of 2 and 3 years
  BMI in kg/m2
morbidity data | between 2 and 3 years of age
  number of morbidity episodes
development | at 2 and 3 years of age
  developmental assessment via Bayley-4

CONTACTS AND LOCATIONS:
Overall Officials: Yannis Manios, Prof, Principal Investigator — Harokopio University
Locations (3):
- Greece (3):
  - Harokopio University, Athens
  - International Hellenic University, Thessaloniki
  - University of Thessaly, Trikala

IPD SHARING:
Plan to Share IPD: No